CLINICAL TRIAL: NCT05553392
Title: StrataXRT Versus Aquaphor for the Prevention and Management of Radiation Dermatitis in Cancer Patients Receiving Elective Inguinal Radiation Therapy
Brief Title: StrataXRT Versus Aquaphor for the Prevention and Management of Radiation Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol deviations and slow recruitment
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SPASX018
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- StrataXRT (Experimental): Studied products will be applied as per the patient information leaflet following manufacturer guidelines to the treatment area. The studied products will be used starting on the first day of radiation therapy. The studied products will be applied twice a day to both the right and left inguinal regions. The studied products will be used daily during the entire course of radiotherapy including on weekends and holidays until at least 4 weeks upon completion of radiation therapy or otherwise until resolution of RD on both sides.
  Interventions: Device: StrataXRT
- Aquaphor (Active Comparator): Studied products will be applied as per the patient information leaflet following manufacturer guidelines to the treatment area. The studied products will be used starting on the first day of radiation therapy. The studied products will be applied twice a day to the entire treatment field. The studied products will be used during the entire course of radiotherapy and for a further 4 weeks upon completion of radiation therapy.
  Interventions: Drug: Aquaphor

INTERVENTIONS:
Device: StrataXRT — StrataXRT is a full contact flexible wound dressing for the prevention and treatment of radiation dermatitis. StrataXRT is a semi-occlusive, self-drying and transparent gel.
  When used as directed StrataXRT dries to form a protective layer that is gas permeable and waterproof which hydrates and protects compromised skin areas and superficial wounds from chemical and microbial invasion. StrataXRT may be directly applied to radiation dermatitis, compromised skin surfaces, superficial wounds and first and second degree burns.
  Arms: StrataXRT
Drug: Aquaphor — Aquaphor is a brand of over-the-counter (OTC) skin care ointments manufactured by Beiersdorf Inc.
  Aquaphor contains 41 percent petrolatum (or petroleum jelly), the active ingredient, temporarily protects minor cuts, scrapes, and burns; protects and helps relieve chapped or cracked skin and lips; helps protect from the drying effects of wind and cold weather.
  Arms: Aquaphor

SUMMARY:
The aim of this study is to assess the efficacy and safety of StrataXRT® in comparison to standard of care (defined using the Common Terminology Criteria for Adverse Events [CTCAE], version 5.0) by assessing the severity of inguinal RD in patients receiving elective radiation therapy +/- systemic therapy to the bilateral inguinal nodes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy of at least 6 months
* Biopsy-confirmed malignancy without gross nodal involvement of the right or left inguinal regions
* Patients will receive elective radiation therapy to bilateral inguinal nodal regions prescribed to 45-50 Gy in 1.8-2 Gy fractions using photon or proton therapy
* No known allergy to studied products
* Able to give written informed consent, or have written consent given on their behalf
* Patients who are able and willing to attend the post-radiation weekly skin assessment appointments
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Abstinence is acceptable if preferred by patient. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Exclusion Criteria:

* Patients with gross cancer involvement of either or both inguinal regions.
* Patients who have received prior pelvic and/or inguinal radiation therapy.
* Patients who cannot apply the studied products to the inguinal region or have it administered to them as required by this study.
* Patients with any medical condition such as active connective tissue disorder that predisposes them to an increased risk of potentially severe radiation dermatitis.
* Patients with existing rashes or wounds in either inguinal region at baseline.
* Planned inguinal dissection within 90 days after completion of radiation therapy on this study.
* Female patients who are pregnant or breast feeding.
* Patients who are unable to give written informed consent, or are unable to have written consent given on their behalf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of acute >grade 2 radiation dermatitis | Until 8 weeks post radiation therapy; up to 4 months
  The Common Terminology Criteria for Adverse Events (CTCAE- Version 5.0) will be used to assess the severity of RD (19). This instrument is routinely used and well validated in radiation oncology for assessing radiation dermatitis (20). This weekly assessment will be undertaken by the assessor who is blinded to the allocation. The assessor will be instructed prior to the first fraction of radiation therapy to score the worst toxicity present, at the time of assessment within the treatment field which consists of the bilateral inguinal regions.
  The amount of > grade 2 RD cases will be compared in both study groups.

SECONDARY OUTCOMES:
Average toxicity assessed using the CTCAE | Until 8 weeks post radiation therapy; up to 4 months
  The Common Terminology Criteria for Adverse Events (CTCAE- Version 5.0) will be used to assess the severity of RD. Patients will be assessed in a repeated measurement model following the visits calendar. The assessments will be pooled based on their visit week and cumulative dose.
  The repeated measurements average toxicity will be compared in both study groups.
Time to onset of moist desquamation | Until 8 weeks post radiation therapy; up to 4 months
  The Common Terminology Criteria for Adverse Events (CTCAE- Version 5.0) will be used to assess the severity of RD.Patients will be assessed in a repeated measurement model following the visits calendar. The assessments will be pooled based on their visit week and cumulative dose.
  The time to moist desquamation will be compared in both study groups.
Pain scores | Until 8 weeks post radiation therapy; up to 4 months
  The participant will be asked to rate their pain level at the irradiated area. The time of interest of the original VAS is modified from "the past 24 hours" to "the past 7 days" for the specific purpose of this study. The VAS has been selected as it is a brief and easy tool for the assessment of pain within both the clinical and research settings. It has been well validated in both the chronic pain and cancer settings. The scale of 0 to 10 is simple for patients to use and reflects common clinical assessment of pain.
  Patients will be assessed in a repeated measurement model following the visits calendar. The assessments will be pooled based on their visit week and cumulative dose.
  The average pain will be compared in both study groups. The worst pain will be compared in both study groups. Pain relief will be measured in the repeated measurements analysis.
Itchiness score | Until 8 weeks post radiation therapy; up to 4 months
  Itching will be scored on a numeric analogue scale of 0-10 in the treated skin (0= no itching at all), (10= itching as bad as you can imagine). Patients will be assessed in a repeated measurement model following the visits calendar. The assessments will be pooled based on their visit week and cumulative dose.
  The average pain will be compared in both study groups. The worst pain will be compared in both study groups. Pain relief will be measured in the repeated measurements analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Cancer Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No